CLINICAL TRIAL: NCT06872840
Title: Addressing Fear of Cancer Recurrence in Parents of Pediatric Cancer Survivors: Adapting The Fear Of Recurrence Therapy (FORT) for Parents and Establishing Acceptability and Feasibility
Brief Title: Adapting The Fear Of Recurrence Therapy (FORT) for Parents and Establishing Acceptability and Feasibility
Acronym: Parent-FORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Sophie Lebel, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-08-24-10241; 506459 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-03-01; First posted 2025-03-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Parent; Fear of Cancer Recurrence; CBT; Childhood Cancer Survivors
Keywords: Pilot study; Group Therapy; Virtual
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT/Existential Group Therapy for Fear of Cancer Recurrence (Experimental): Participants will receive 7 weekly group therapy sessions consisting of psychoeducation on fear of cancer recurrence, relaxation training, CBT, and evidenced-based tips to decrease avoidance and anxiety surrounding fear of cancer recurrence.
  Interventions: Behavioral: Parent Fear of Recurrence Therapy (Parent-FORT)
- Waitlist Control Group (No Intervention): Participants assigned to this arm will wait about 3-months to receive the intervention.

INTERVENTIONS:
Behavioral: Parent Fear of Recurrence Therapy (Parent-FORT) — 7 weekly sessions of 120 minutes each. During the 7 weeks, participants will be asked to participate in activities, participate in group discussions, and complete homework assignments.
  Arms: CBT/Existential Group Therapy for Fear of Cancer Recurrence

SUMMARY:
Clinical levels of fear of cancer recurrence (FCR) affect up to 59% of adult cancer survivors. Family caregivers experience equal or greater levels of FCR, which has been linked to lower quality of life and increased distress. FCR can be addressed in cancer survivors with brief interventions. However, none of these interventions have been tested with parents of childhood cancer survivors. This is an urgent gap: the survival rates of childhood cancer have increased more rapidly than for adult cancers, resulting in a growing population of childhood cancer survivors who, along with their families, need support.

The goals of this pilot study are to demonstrate 1) that a newly adapted intervention of FORT (Parent-FORT) is feasible (i.e., participant recruitment, attendance and participation) and acceptable (i.e., parent satisfaction of the intervention) for a larger study, and 2) the clinical implications of Parent-FORT on fear of cancer recurrence (FCR) and quality of life in parents of childhood cancer survivors.

Parents will be randomly assigned to participate in the Parent-FORT intervention immediately or a three-month waitlist control group. They will complete a questionnaire package before and after the intervention, as well as at a three month follow up. This study will help bridge an important gap in bringing evidence-based care to parents who have never been offered help before for their FCR.

DETAILED DESCRIPTION:
Pilot Study:

36 parents will be recruited to participate in the study. Additionally, 3 therapists with extensive online support group experience to conduct the Parent-FORT videoconference therapy sessions. Therapist competency to administer Parent-FORT will be determined by registered professionals in counselling or psychotherapy, experience in psychosocial oncology, specifically with parents, and having led at least one group. Interested parents will contact the research coordinator, via telephone or email, to be screened for eligibility and to complete the consent forms. This pilot study will serve as a first step in potential sample size calculations and recruitment times. For this pilot study, active recruitment will last for a period of 15 months during which 36 parents are aimed to be recruited in order to create 4 groups of 9 participants (2 intervention conditions and 2 WLCG). Feasibility of recruitment for the larger RCT will be determined using these criteria: 1) If during our recruitment period less than 18 participants, recruitment for a larger RCT, using our current recruitment strategies, will be deemed not feasible, 2) If between 18 and 25 participants are recruited, then a larger multicentre approach for recruitment will be considered, 3) If recruit 25 participants or more, recruitment for a larger RCT, using our current methods, will be deemed feasible. The sample size will be reevaluated for the larger RCT based on the results from this pilot study.

Parent-FORT consists of 7 consecutive weekly group sessions of 120 minutes each offered through videoconference and weekly assigned homework. Parent-FORT is therapist led, however participants will receive a workbook where they can follow along, take notes, and complete the exercises and the homework assignments. The overall aim of Parent-FORT is to guide Parent towards a more manageable level of worry and fear of recurrence. The key goals are to: 1) distinguish worrisome symptoms from benign ones; 2) identify FCR triggers and inappropriate coping strategies; 3) facilitate the learning and use of new coping strategies, such as relaxation techniques, cognitive restructuring, communication strategies and the use of self-care; 4) increase tolerance for uncertainty; 5) promote emotional expression of specific fears that underlie FCR; and 6) re-examine life priorities and set realistic goals for the future. Each session is composed of exercises where participants have to answer questions, share with the group or watch videos. Furthermore, homework is assigned after each session to be completed before next week's session. Eligible participants will attend a one-on-one pre-therapy meeting with a study therapist to prepare them for the group work (i.e.: review expectations and assess whether group work is appropriate for the participant) and complete the 7-week Parent-FORT intervention. Membership will be closed once groups are formed and the sessions have started to enhance group cohesiveness and consistency. Before starting the intervention, participants will receive a standardized manual describing each session's activities and assignments. All participants (including those in the wait list control group) will complete a questionnaire package pre intervention, post intervention, and at a three month follow up via Qualtrics. Additionally, participants will be asked to complete post session measures, namely the Working Alliance Inventory - Revised Short Form as well as the Group Cohesiveness Scale after the 1st, 4th and 7th sessions.

Therapist Training and Supervision:

To enhance therapist adherence to treatment, the therapists recruited for the study will be provided with a standardized Parent-FORT manual and will be trained by the research psychologists through an online training. The research team will review the video of each session, and the principal investigator will provide weekly 30-minute supervision to the therapists. Furthermore, the study will use an updated version of the fidelity checklist that was used to evaluate adherence during the previous FORT studies. If adherence is less than 80% on any session, the research team will provide additional over-the-telephone feedback to the therapists running the group. This approach to monitoring treatment integrity and fidelity has been successful in previous FORT studies.

Qualitative Assessment:

To gain further insights about the feasibility, acceptability, and potential clinical significance of Parent-FORT, all study participants will be asked to complete semi-structured exit interviews. This will enable a holistic understanding of their experience of Parent-FORT, elucidate key intervention processes, and identify additional secondary outcomes. Lastly, the research coordinator will attempt to interview participants who dropped out of the intervention, to understand any hindering factors. Consenting participants will be asked to complete a semi structured interview (30-60 minutes) about their experience of the intervention through videoconferencing.

Randomization:

This study will use a mixed method randomized control trial design using a waitlist control group and 3 months follow up, with 18 participants per condition. To minimize attrition associated with waiting to enroll participants, block randomization will be used. Specifically, a list of 4 blocks with equal numbers of intervention (I) and wait list control (WLCG) groups (e.g. I-I-WLCG-WLCG; I-WLCG-WLCG-I, etc.) will be randomly created. Once the first 9 participants have been recruited, they will be assigned to whichever group came up first on the list. The next 9 participants will be assigned to the next group on the generated list until all 4 groups have been completed. Participants assigned to the WLCG will be offered the intervention after the 3-month period. To limit bias, each of the 4 blocks of the list will be in separate sealed envelopes that will be opened one at a time after 9 participants have been recruited.

Minimizing Dropouts and Attrition:

To maximize attendance, as in our prior research, participants will be told during informed consent procedures about the importance of attending all 7 sessions to ensure benefit from the intervention. Participants will receive two email reminders about each upcoming session, along with "homework" and session pre-reading materials. They will be asked to inform group therapists if they are to be absent. For participants who miss a session, they will be offered one individual videoconference make-up session for their first missed session before the next group; they will not be offered subsequent make-up sessions for additional missed sessions to decrease the risk that this would encourage those who prefer individualized attention to miss group sessions. Participants who miss more than two sessions will be asked to stop the intervention and restart with the next available group. This approach was successfully tested in previous FORT studies. To minimize differential attrition from the WLCG participants, participants will be emailed monthly with an update about the wait time.

Feasibility and Acceptability Criteria:

The following criteria will be used to assess the feasibility and acceptability of Parent-FORT: 1) ability to recruit 36 parents in 15 months; 2) ability to randomize these 36 parents; 3) ability to deliver Parent-FORT to 27 Parent in 15 months (25% dropout rate); 4) 80% completion of 6 out of the 7 sessions; 5) complete measures for 90% of participants; 6) ability to deliver Parent-FORT as intended as measured by a fidelity rating of above 80% on 75% of reviewed sessions; and 7) Parent satisfactory ratings >than 80% in terms of its content, therapists, and mode of delivery.

Quantitative analysis:

Descriptive statistics will be used to report on FCR outcomes. A linear mixed-effect model analyses will be done on the secondary outcome measures pre- and post-intervention and at the 3-month follow-up. All analyses will use both an intent-to-treat and per protocol approaches. Known extraneous variables that could influence FCR (e.g., age, education, income, cancer stage) will be measured and control for, and monitor for participants' use of any additional psychological support at each data-collection time-points. Dependence of the group data will be analyzed with an intraclass correlation coefficient (p) using a multilevel model.

Qualitative Analysis:

Conventional content analysis will be used to analyse the qualitative data. Interviews will be audiotaped, transcribed verbatim, and managed using the qualitative software program NVivo. Transcripts will be systematically coded into anticipated (e.g., motivations to participate, benefits of participation) and emergent codes. This is an iterative process whereby an initial set of themes are coded, applied to new transcripts, and revised to adjust for new information, until no new codes emerge. Double coding of 80% of the interviews will be done by the research assistant. These codes will then be sorted into subcategories (ideally between 10 to 15).

ELIGIBILITY:
Inclusion Criteria:

* Parent (or primary caregiver) caring for a childhood cancer survivor (<18 years of age) of any type of cancer type, who is at least 1 months from the completion of active treatment and has not had a recurrence of their cancer
* A score of 13 or greater on the Fear of Cancer Recurrence Inventory-Short Form-Parent version (FCRI-SF-P; range 0-36), suggesting clinical levels of FCR
* Access to a computer and internet connection
* Living in Canada

Exclusion Criteria:

* Being the parent of a pediatric cancer survivor who is now 18 years of age or older
* Being the parent of a pediatric cancer survivor who has undergone hematopoietic cell transplantation and has active chronic or acute graft-versus-host disease which has not stabilized for at least 3 months
* Non-English speakers
* Currently participating in another therapist-led psychosocial therapy group
* Parent with unmanaged/undermanaged mental health disorder judged to be clinically contraindicated and/or likely to affect the group work
* To avoid violating the assumption of nonindependence of the data, only one parent/caregiver per child can participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2027-05-26 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline fear of cancer recurrence after intervention | Changes in baseline fear of cancer recurrence 7 weeks after the start of the intervention
  Fear of Cancer Recurrence Inventory - Parent (FCRI-P), range from 0-36 with higher scores indicating high levels of fear of cancer recurrence
Changes in baseline fear of cancer recurrence at three months | Changes in baseline fear of cancer recurrence 3 months after the start of the intervention
  Fear of Cancer Recurrence Inventory - Parent (FCRI-P), range from 0-36 with higher scores indicating high levels of fear of cancer recurrence

SECONDARY OUTCOMES:
Changes in Baseline Intolerance of Uncertainty Scale at 7 Weeks | Changes in baseline Intolerance of Uncertainty Scale after 7 weeks of the intervention
  Intolerance of Uncertainty Scale - Short Form (IUS-SF), range from 12-60 with higher scores indicating high levels of intolerance of uncertainty
Changes in Baseline Intolerance of Uncertainty Scale at 3 Months | Changes in baseline Intolerance of Uncertainty Scale at 3 month after the completion of the intervention
  Intolerance of Uncertainty Scale - Short Form (IUS-SF), range from 12-60 with higher scores indicating high levels of intolerance of uncertainty
Changes in baseline Uncertainty in Illness at 7 weeks | Changes in baseline Intolerance of Uncertainty Scale after 7 weeks of the intervention
  Mishel Uncertainty in Illness Scale Short-Form (MUIS-SF), range from 5-25 with higher scores indicating high levels of uncertainty in illness
Changes in baseline Uncertainty in Illness at 3 months | Changes in baseline Intolerance of Uncertainty Scale at 3 month after the completion of the intervention
  Mishel Uncertainty in Illness Scale Short-Form (MUIS-SF), range from 5-25 with higher scores indicating high levels of uncertainty in illness
Changes in baseline Positive Beliefs About Worrying at 7 weeks | Changes in baseline Positive Beliefs About Worrying after 7 weeks of the intervention
  Why do people Worry about Health Questionnaire (WW-H), range from 13-65 with higher scores indicating more positive beliefs about worrying
Changes in baseline Positive Beliefs About Worrying at 3 months | Changes in baseline Positive Beliefs About Worrying at 3 month after the completion of the intervention
  Why do people Worry about Health Questionnaire (WW-H), range from 13-65 with higher scores indicating more positive beliefs about worrying
Changes in baseline avoidance at 7 weeks | Changes in baseline avoidance after 7 weeks of the intervention
  Cognitive Avoidance Questionnaire (CAQ), range from 25-125 with higher scores indicating higher use of avoidance as a coping strategy
Changes in baseline avoidance at 3 months | Changes in baseline Avoidance at 3 month after the completion of the intervention
  Cognitive Avoidance Questionnaire (CAQ), range from 25-125 with higher scores indicating higher use of avoidance as a coping strategy
Changes in fear of bodily threat at 7 weeks | Changes in fear of bodily threat after 7 weeks of the intervention
  Bodily Threat Inventory-Parent (BTI-Parent), range from 30-150 with higher scores indicating higher levels of fear
Changes in fear of bodily threat at 3 months | Changes in fear of bodily threat at 3 month after the completion of the intervention
  Bodily Threat Inventory-Parent (BTI-Parent), range from 30-150 with higher scores indicating higher levels of fear
Changes in healthcare utilization at 3 months | Changes in healthcare utilization at 3 month after the completion of the intervention
  Healthcare Utilization Questionnaire. Parents will report on the number of times in the past 3 months that they used medical services for their child
Changes in quality of life at 7 weeks | Changes in quality of life after 7 weeks of the intervention
  The EuroQol Five Dimensional Questionnaire (EQ-5D) is a 5-item quality of life measure. Score from 1-5 in each dimension. Higher scores indicates lower quality of life.
Changes in quality of life at 3 months | Changes in quality of life at 3 month after the completion of the intervention
  The EuroQol Five Dimensional Questionnaire (EQ-5D) is a 5-item quality of life measure (EQ-5D). Score from 1-5 in each dimension. Higher score indicates lower quality of life.
Changes in perceived risk of recurrence at 7 weeks | Changes in perceived risk of recurrence after 7 weeks of the intervention
  Perceived risk of recurrence will be assessed using a one-item question
Changes in perceived risk of recurrence at 3 months | Changes in perceived risk of recurrence 3 month after the completion of the intervention
  Perceived risk of recurrence will be assessed using a one-item question
Measure of acceptability/satisfaction at 7 weeks | Measure of acceptability/satisfaction after 7 weeks of the intervention
  Treatment Acceptability and Preferences (TAP) measure, range from 4-20, with higher scores indicating greater acceptability/satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lebel, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamarche J, Nissim R, Avery J, Wong J, Maheu C, Lambert SD, Laizner AM, Jones J, Esplen MJ, Lebel S. It is Time to Address Fear of Cancer Recurrence in Family Caregivers: Feasibility and Acceptability of a Randomized Pilot Study of the Family Caregiver Version of the Fear of Recurrence Therapy (FC-FORT). Psychooncology. 2025 Feb;34(2):e70084. doi: 10.1002/pon.70084. PMID 39887474
- [Background] Murphy LK, Heathcote LC, Prussien KV, Rodriguez EM, Hewitt JA, Schwartz LE, Ferrante AC, Gerhardt CA, Vannatta K, Compas BE. Mother-child communication about possible cancer recurrence during childhood cancer survivorship. Psychooncology. 2021 Apr;30(4):536-545. doi: 10.1002/pon.5600. Epub 2020 Dec 3. PMID 33227159
- [Background] Webb K, Sharpe L, Butow P, Dhillon H, Zachariae R, Tauber NM, O'Toole MS, Shaw J. Caregiver fear of cancer recurrence: A systematic review and meta-analysis of quantitative studies. Psychooncology. 2023 Aug;32(8):1173-1191. doi: 10.1002/pon.6176. Epub 2023 Jun 11. PMID 37303263
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Lebel S, Ozakinci G, Humphris G, Mutsaers B, Thewes B, Prins J, Dinkel A, Butow P; University of Ottawa Fear of Cancer Recurrence Colloquium attendees. From normal response to clinical problem: definition and clinical features of fear of cancer recurrence. Support Care Cancer. 2016 Aug;24(8):3265-8. doi: 10.1007/s00520-016-3272-5. Epub 2016 May 12. PMID 27169703
- See also: Related Info — https://www.psolab.ca/research/parent-fort